CLINICAL TRIAL: NCT00051493
Title: ALIMTA Plus Carboplatin as Front-Line Chemotherapy for Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer: A Phase 2 Clinical Trial.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6142; H3E-MC-JMEZ
Record Dates: First submitted 2003-01-10; First posted 2003-01-14 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; NSCLC; Advanced Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed; Carboplatin

INTERVENTIONS:
Drug: ALIMTA
Drug: Carboplatin

SUMMARY:
The purpose of this study is to evaluate the effects (good and bad) of LY231514 (ALIMTA) and Carboplatin on you and your non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* You have a diagnosis of non-small cell lung cancer.
* You have received no prior chemotherapy.
* You have at least one measurable lesion.
* You have an adequate performance status.
* You are at least 18 years of age.

Exclusion Criteria:

* You have previously received chemotherapy for your lung cancer.
* You have received radiation within the last 30 days.
* You have active infection or other serious condition.
* You have brain metastasis.
* You have recently lost a significant amount of weight.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-04; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Locations (1):
- Houston, Texas, United States